CLINICAL TRIAL: NCT05029895
Title: A Post-Marketing Observational Study to Evaluate Safety and Effectiveness of Upadacitinib in Adolescent Patients Ages 12 to <18 Years Old Diagnosed With Atopic Dermatitis (AD)
Brief Title: A Study to Evaluate Adverse Events and Change in Disease State of Oral Upadacitinib in Adolescent Participants Ages 12 to <18 Years Old Diagnosed With Atopic Dermatitis (AD)
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-442
Record Dates: First submitted 2021-08-30; First posted 2021-09-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Atopic Eczema; Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving upadacitinib for atopic dermatitis.

SUMMARY:
Atopic dermatitis (AD; also known as atopic eczema) is an inflammatory skin disease. The safety and effectiveness of upadacitinib for AD has been well-documented in previous studies, however, these studies included a limited number of adolescent patients in Japan. Therefore, the purpose of this observational study is to evaluate safety and effectiveness of upadacitinib in adolescent AD participants age 12 to <18 years old in Japan in the real-world setting.

Upadacitinib is an approved drug being developed for the treatment of AD in adolescents in Japan. Around 170 participants age 12 to <18 who are prescribed upadacitinib for the treatment of AD in routine clinical practice will be enrolled at multiple sites in Japan.

Participants will receive oral upadacitinib as prescribed by their physician. Data from these participants will be collected for approximately 2 years.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the course of the study at a hospital or clinic and will be asked to provide additional information by questionnaire at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are diagnosed with atopic dermatitis (AD).
* History of topical anti-inflammatory agents such as topical steroids and topical tacrolimus for AD.
* Participants initiating upadacitinib for the treatment of AD in routine clinical practice.
* Body weight >=30 kg at the start of dosing.

Exclusion Criteria:

* Prior treatment with upadacitinib
* Currently participating in another registrational clinical research study
* Participants for whom upadacitinib is contraindicated

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent participants receiving upadacitinib according to the product prescribing information for atopic dermatitis in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Infection | 2 Years
  Serious infection is defined as any infection identified as an Infection Company MedDRA Query that meets seriousness criteria

SECONDARY OUTCOMES:
Percentage of Participants Reporting an Adverse Event (AE)/Adverse Drug Reaction (ADR) including Safety Specification | 2 Years
  An AE/ADR is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. Safety specification is defined as: serious infections (including TB, pneumonia, pneumocystis pneumonia, pulmonary hemorrhage and opportunistic infections), herpes zoster, VTE (deep venous thrombosis and pulmonary embolus), gastrointestinal perforation, hepatic function disorder, Interstitial lung disease, neutrophil count decreased, lymphocyte count decreased and hemoglobin decreased, hepatitis B virus reactivation, malignancies, major adverse cardiac events, rhabdomyolysis and myopathy, and renal impairment, and safety in pediatric patients and weighing <40 kg.
Percentage of Participants Reporting an Adverse Event (AE)/Adverse Drug Reaction (ADR) Related to Impact on Bone Growth | 2 Years
  An AE/ADR is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious AE (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent AEs/treatment-emergent SAEs (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vlGA-AD) of 0 or 1 | 2 Years
  The vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).
Absolute Change from Baseline in Worst Pruritus-Numeric Rating Scale (NRS) | Up to 2 Years
  Worst Pruritus NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percent Change from Baseline in Worst Pruritus-Numeric Rating Scale (NRS) | Up to 2 Years
  Worst Pruritus NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving an Improvement in Worst Pruritus-NRS >=4 | 2 Years
  Worst Pruritus NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Percentage of Participants Achieving Worst Pruritus-NRS 0/1 | 2 Years
  Worst Pruritus NRS is a validated single self-reported item designed to measure peak pruritus, or 'worst' itch, over the previous 24 hours with a higher score denoting worse itch.
Absolute Change from Baseline in Patient Oriented Eczema Measure (POEM) Score | 2 Years
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale with a higher score denoting worse AD.
Percent Change from Baseline in POEM Score | 2 Years
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale with a higher score denoting worse AD.
Percentage of Participants Achieving a Clinically Meaningful Improvement in POEM | 2 Years
  The POEM is a 7-item, validated questionnaire used in clinical practice and clinical trials to assess disease symptoms in both children and adults. Subjects respond to 7 items, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale with a higher score denoting worse AD. Minimal Clinically Important Difference=4

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (61):
- Japan (61):
  - Takeo Skin Clinic /ID# 248095, Asahi Owari, Aichi-ken
  - Ichinomiya Municipal Hospital /ID# 245070, Ichinomiya-shi, Aichi-ken
  - NHO Nagoya Medical Center /ID# 245069, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 250809, Nagoya, Aichi-ken
  - Aichi Children's Health and Medical Center /ID# 245357, Obu-shi, Aichi-ken
  - Noriko Dermatology Clinic /ID# 246626, Akita, Akita
  - Nippon Medical Chiba Hokusoh Hospital /ID# 246627, Inzai-shi, Chiba
  - National Hospital Organization Shimoshizu National Hospital /ID# 245064, Yotsukaido-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 248739, Matsuyama, Ehime
  - Aso Iizuka Hospital /ID# 252145, Iizuka-shi, Fukuoka
  - Kurume University Hospital /ID# 248740, Kurume-shi, Fukuoka
  - Hoshi General Hospital /ID# 250959, Koriyama-shi, Fukushima
  - Central Japan International Medical Center /ID# 246625, Minokamo-shi, Gifu
  - Hiroshima University Hospital /ID# 245356, Hiroshima, Hiroshima
  - Kitami Red Cross Hospital /ID# 250838, Kitami-shi, Hokkaido
  - Takagi Dermatological Clinic /ID# 241160, Obihiro-Shi, Hokkaido
  - Hosui General Medical Clinic /ID# 241881, Sapporo, Hokkaido
  - Duplicate_Kobayashi Skin Clinic /ID# 248006, Sapporo, Hokkaido
  - Hayano Pediatrician Clinic /ID# 250960, Himeji-shi, Hyōgo
  - Kobe City Medical Center General Hospital /ID# 244052, Kobe, Hyōgo
  - Kobe City Medical Center General Hospital /ID# 250836, Kobe, Hyōgo
  - Bito Dermatology Clinic /ID# 244093, Kobe, Hyōgo
  - Maekawa Kids Clinic /ID# 249521, Sichuan, Hyōgo
  - Mito Kyodo General Hospital /ID# 243745, Mito, Ibaraki
  - Torii Dermatology Clinic /ID# 252143, Nonoichi-shi, Ishikawa-ken
  - Takeoka Dermatology Clinic /ID# 240610, Marugame, Kagawa-ken
  - Kagoshima City Hospital /ID# 252142, Kagoshima, Kagoshima-ken
  - Imamura General Hospital /ID# 249526, Kagoshima, Kagoshima-ken
  - Kagoshima University Hospital /ID# 248732, Kagoshima, Kagoshima-ken
  - Hiratsuka City Hospital /ID# 245071, Hiratsuka-shi, Kanagawa
  - Teikyo University Mizonokuchi Hospital /ID# 252146, Kawasaki, Kanagawa
  - National Hospital Organization Sagamihara National Hospital /ID# 243744, Sagamihara-shi, Kanagawa
  - Kanagawa Children's Medical Center /ID# 252144, Yokohama, Kanagawa
  - National Mie Hospital /ID# 245066, Tsu, Mie-ken
  - Okayama University Hospital /ID# 252141, Okayama, Okayama-ken
  - Naha City Hospital /ID# 245065, Naha, Okinawa
  - Kansai Medical University Hospital /ID# 246020, Hirakata-shi, Osaka
  - Kansai Medical University Takii Hospital /ID# 250195, Moriguchi, Osaka
  - Duplicate_Japanese Red Cross Osaka Hospital /ID# 249524, Osaka, Osaka
  - Osaka Metropolitan University Hospital /ID# 245972, Osaka, Osaka
  - Hino Clinic /ID# 245975, Sakai-shi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital /ID# 251660, Takatsuki-shi, Osaka
  - Okada Kodomonomori Clinic /ID# 248096, Kasukabe-shi, Saitama
  - Saitama Medical Center /ID# 244695, Kawagoe, Saitama
  - Dokkyo Medical University Saitama Medical Center /ID# 249525, Koshigaya, Saitama
  - Nagahama Red Cross Hospital /ID# 252136, Nagahama-shi, Shiga
  - Shiga University of Medical Science Hospital /ID# 245969, Ōtsu, Shiga
  - Chutoen General Medical Center /Id# 248741, Kakegawa-shi, Shizuoka
  - Chutoen General Medical Center /Id# 249522, Kakegawa-shi, Shizuoka
  - Dokkyo Medical University Hospital /ID# 245068, Mibu, Tochigi
  - Tokyo Med Univ Hachioji Med Ct /ID# 250958, Hachioji-shi, Tokyo
  - National Center For Child Health And Development /ID# 244696, Setagaya City, Tokyo
  - Tokyo Metropolitan Hiroo Hospital /ID# 250837, Shibuya Ward, Tokyo
  - Fraternity Memorial Hospital /ID# 245974, Sumida-ku, Tokyo
  - Sugamo Sengoku Dermatology /ID# 247761, Toshima City, Tokyo
  - Tonami General Hospital /ID# 247760, Tonami-shi, Toyama
  - Suzuki Kids Clinic /ID# 243743, Shingū, Wakayama
  - Wakayama Medical University Hospital /ID# 247498, Wakayama, Wakayama
  - Yamaguchi Grand Medical Center /ID# 251659, Hohu-shi, Yamaguchi
  - Fukuoka Children'S Hospital /ID# 245067, Fukuoka
  - Takatsuki General Hospital /ID# 242334, Osaka

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/